CLINICAL TRIAL: NCT00081861
Title: A Phase II Study of Avastin Plus Rituximab for Patients With Relapsed and Chemotherapy- or Rituxan-Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma
Brief Title: Avastin Plus Rituximab for Patients With B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0520
Record Dates: First submitted 2004-04-23; First posted 2004-04-27 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Lymphoma
Keywords: Non-Hodgkin's Lymphoma; B-Cell Lymphoma; Lymphoma; Avastin; Bevacizumab; Rituximab; Rituxan
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Bevacizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin + Rituximab (Experimental): Avastin 10 mg/kg given intravenously every 2 weeks for 4 doses, and Rituximab 375 mg/m^2 intravenously weekly for 8 doses.
  Interventions: Drug: Avastin; Drug: Rituximab

INTERVENTIONS:
Drug: Avastin — 10 mg/kg given intravenously every 2 weeks for 4 doses.
  Other Names: Bevacizumab
Drug: Rituximab — 375 mg/m^2 given intravenously weekly for 8 doses, 30 minutes to 1 hour following Bevacizumab.
  Other Names: Rituxan

SUMMARY:
Phase II Study of Avastin Plus Rituximab for Patients with Relapsed and Chemotherapy - or Rituxan Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
Bevacizumab is a new research drug that may help to stop or slow the growth of blood vessels in your tumor. These blood vessels are needed by the tumor to grow. Rituxan is a commercially available drug that is commonly used to treat relapsed and refractory lymphoma.

Before treatment starts, you will be asked questions about your medical history and about any surgeries you have had. You will have a complete physical exam including blood (around 3 tablespoons) and urine tests. You will have a sample of bone marrow collected to learn if the lymphoma has spread to the bone marrow. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. You will have either a CT scan or a MRI of the neck, chest, abdomen, and pelvis, and you will have a gallium or PET scan. You will be asked about any medications that you are taking, including over-the-counter medications. Women who are able to have children must have a negative blood pregnancy test.

Additional blood samples (2 tablespoons) will be collected from you before starting therapy and every 2 months during this study for tests to help your doctors and researchers to learn more about how Bevacizumab works.

During the study, you will be given a dose of rituximab by vein once a week for 8 weeks in a row, and a dose of Bevacizumab every other week. The drugs will be contained in a bag and will be given to you through a needle in one of your veins. This method of giving the drugs is called an infusion. The infusion of Bevacizumab may take 1 to 2 hours, and the infusion of rituximab may take up to 3 to 6 hours. This method of giving a drug is called an infusion. In the first week, infusions of rituxan and Bevacizumab will be given on the same day.

During the infusion of each drug, you will have your vital signs checked often and you will be watched for any side effects. If you experience side effects, the infusion may be slowed down or stopped until the symptoms have gone away.

Within 2 weeks after your 8th dose of rituximab, (4th dose of Bevacizumab) you will have a follow-up visit scheduled to evaluate the status of the disease. During the follow-up visit, you will have a physical exam and blood (around 4 tablespoons) will be collected for lab tests. You will have a CT scan or a MRI, gallium or PET scan, and bone marrow biopsy (if needed). If the disease gets worse or you experience any intolerable side effects, you will be taken off the study. If you are taken off the study or your doctor decides that you should stop study treatment, you will be asked to return to M. D. Anderson for all of the scheduled follow-up visits to check for long term side effects of the drug and to check on the status of the disease.

If the disease remains stable or shrinks after 8 weeks of therapy, you may continue to receive Bevacizumab treatments every 2 weeks for a maximum of a total of 6 months. Even if the treatment is shown to be of benefit to you, your doctor may not continue to give you additional treatments with Bevacizumab beyond the total of 6 months.

After treatment, you will have follow-up visits scheduled to check on the status of the disease. These visits will be scheduled every 3 months for 1 year, then every 4 months for 1 more year, then every 6 months until the disease gets worse. During these visits, you will have a physical exam, blood tests (around 2 tablespoons), and either a CT scan or a MRI. You will also have a sample of bone marrow collected.

This is an investigational study. Bevacizumab has been authorized by the FDA for use in research only. Rituximab is FDA approved and is commercially available. There will be no cost for Bevacizumab or for any tests and procedures that are not considered part of standard of care. Up to 40 patients will take part in this study. All patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Must have bi-dimensionally measurable, recurrent or chemotherapy - or Rituxan-refractory aggressive B-cell NHL (Diffuse large B-cell, transformed B-cell lymphoma, or Mantle cell lymphoma)
* Patient who relapse after autologous (not allogeneic) stem cell transplantation are eligible.
* Patients must have had prior Rituximab therapy, with response duration of at least 6 months to the last Rituximab-based therapy (single agent or in combination)
* No anti-lymphoma therapy within the past 3 weeks, and no radiation therapy within 2 weeks.
* Patients must not be eligible for treatment of a higher priority.
* Must have a good performance status (<3 Zubrod, >/=60 Karnofsky).
* Must have a good marrow reserve: ANC >/=1,000, Platelets >/=75,000.
* Bilirubin </= 2mg/dl, SGOT or SGPT </= x 5 normal values.
* Age > 18 (There is no information about the toxicity of Bevacizumab especially adverse effects on growth and development in pediatric patients).
* Must sign a consent form.
* Must have a life expectancy of > 12 weeks.

Exclusion Criteria:

* HIV positive
* History of serious cardiac disease such as myocardial infarction within 6 months of treatment, brady- or tachyarrhythmia, or clinically uncontrolled hypertension (blood pressure >160/110 mmHg).
* Active infection or history of opportunistic infection.
* Pregnant women or breast-feeding women.
* Women of child-bearing age who are not practicing adequate contraception.
* History of prior DVT or pulmonary embolus.
* INR > 1.5
* Serum creatinine > 2mg/dl, or clinically significant proteinuria (patients with >1+ proteinuria should have 24 hour urine collection and those with >2gm/day should be excluded).
* Evidence of bleeding diathesis or coagulopathy.
* History of other cancers within 5 years except for basal cell carcinoma of the skin.
* Radiotherapy within 14 days of Day 0.
* Current, recent (within 21 days of Day 0), or planned participation in an experimental drug study.
* Hemoglobin <9gm/dl (may be transfused or receive epoetin alfa [e.g., Epogen]to maintain or exceed this level).
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of CNS disease (including CNS involvement from primary cancer) or hemorrhagic or thrombotic stroke within the last 6 months.
* History of hemoptysis requiring transfusion and/or hospitalization within the last 5 years.
* Anatomic lesion that increase the risk of serious hemorrhage (e.g., invasion of a major vessel by tumor).
* Current, ongoing treatment with full-dose warfarin or its equivalent.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0.
* Fine needle aspirations, indwelling catheter placement, or core biopsy within 7 days prior to Day 0.
* Anticipation of need for major surgical procedure during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pro, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2004 through November 2006. All participants recruited at U.T. M.D. Anderson Cancer Center.
Period: Overall Study
Arm/Group | Avastin + Rituximab
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avastin + Rituximab
Number analyzed (Participants) | 13
Age Continuous [Median (Full Range); unit: years] | 67 [34 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response (Complete Response or Progressive Disease)
Description: Response criteria according to the International Working Group Recommendations for lymphoma where Complete Response (CR) defined as "complete disappearance" of clinically detectable disease and Progressive Disease defined by disease appearance by complete blood count (CBC), clinical and radiologic findings, and/or sizes of lymph nodes, spleen, and liver. Response measured from first documentation of response to first detection of progression.
Time Frame: After 8 weeks of therapy (4 doses of Avastin and 8 doses of Rituximab),
Population: Two participants received first treatment dose but were not eligible for response.
Measure: Number; unit: Participants
Arm/Group | Avastin + Rituximab
Number analyzed (Participants) | 11
Participants
  Complete Response | 2
  Progressive Disease | 6

ADVERSE EVENTS:
Time Frame: 2 years, 7 months
Arm/Group | Avastin + Rituximab
Serious Adverse Events (participants affected / at risk) | 12/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin + Rituximab (N=13)
Pain (Investigations) | 3 — Abdomen, Chest/Thorax, Head/Headache
Fatigue (General disorders) | 2
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Infection (Infections and infestations) | 4 — Infection with normal or varying Absolute neutrophil count (ANC), Neutrophils, or Platelet levels
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin + Rituximab (N=13)
Diarrhea (Gastrointestinal disorders) | 4
Anemia (Blood and lymphatic system disorders) | 4
Rigors/Chills (Musculoskeletal and connective tissue disorders) | 4
Hypertension (Cardiac disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No